CLINICAL TRIAL: NCT02647801
Title: The SMASH Study: Self-control and Mindfulness Within Ambulatorily Assessed Network Systems Across Health Related Domains
Brief Title: Self-control and Mindfulness Within Ambulatorily Assessed Network Systems Across Health Related Domains
Acronym: SMASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Mario Wenzel, Dipl. Psych. Mario Wenzel, Johannes Gutenberg University Mainz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2015-JGU-psychEK-011
Record Dates: First submitted 2015-12-15; First posted 2016-01-06 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Self Regulation
Keywords: Network approach; mindfulness; self-control; ambulatory assessment
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness intervention (Experimental): The experimental group comes to weekly laboratory meetings and practices mindfulness. Participants also fill out self-report questionnaires which assess self-control and mindfulness.
  Interventions: Behavioral: Mindfulness intervention
- Control group (No Intervention): The control group comes to weekly laboratory meetings and fills out self-report questionnaires which assess self-control and mindfulness. No mindfulness training is carried out.

INTERVENTIONS:
Behavioral: Mindfulness intervention — Mindfulness is practiced with a weekly computer based guided breathing meditation in which one's own breath has to be counted repetitively from 1 to 9. Participants have to press a specific button for breaths 1 to 8 and then press another button for breath 9 on a keyboard. During this practice they put on headphones and listen to a voice that guides them through breathing meditation. A "click" sound will occur if breath is miscounted (Levinson et al., 2014). After each computer based breathing meditation the experimenter and participants exchange meditation experiences and views. After the first mindfulness training participants in the experimental group are also able to practice mindfulness at home by listening to audio files on the mobile phone (bodyscan or breathing meditation).
  Arms: Mindfulness intervention

SUMMARY:
The aim of this trial is to test a novel network approach (Bringmann et al., 2013), which enables to investigate the complex, interdependent network of self-control and its influences in everyday life. By adding an intervention to the network, such as mindfulness training, it is also possible to explore the way mindfulness changes connection strengths between network variables.

For six weeks, an ambulatory assessment and additional seven weekly laboratory sessions are conducted with 120 students from the Johannes Gutenberg University Mainz who are randomized to a control (n=60) or intervention condition (n=60). Pre and post measurement sessions take place to assess self-reported trait self-control and mindfulness and a behavioral measure of mindfulness (Levinson, Stoll, Kindy, Merry & Davidson 2014). Participants of both the experimental and control condition come to five weekly lab meetings in which they fill out questionnaires to assess changes in self-reported self-control and mindfulness. But only participants of the experimental condition take part in weekly computer based mindfulness trainings. During the ambulatory assessment, participants complete questionnaires six times a day via mobile phones that are randomly prompted and answer questions about state self-control, motivation, affect, and current situation.

ELIGIBILITY:
Inclusion Criteria:

* understanding and speaking German
* aged between 18 and 65 years
* knowledge about how to use a mobile phone

Exclusion Criteria:

* psychological disease
* mental or somatic disability that could impair the usage of a mobile phone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 137 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Three items from the State Self-control Capacity Scale (SSCCS) | From day 1 till day 40, six times a day between 10 am and 8 pm
  German version of the SSCCS. Self-report on current self-control capacity of participants.
Three items from the Mindfulness Attention Awareness Scale (MAAS) | From day 1 till day 40, six times a day between 10 am and 8 pm
  Items from the German version of the MAAS. Self-report on current mindfulness of participants.

SECONDARY OUTCOMES:
Eight affect items based on the affective circumplex (Russel, 2003) | From day 1 till day 40, six times a day between 10 am and 8 pm and at weekly laboratory meetings
  Eight items which Kuppens and colleagues used for an experience sampling study (Kuppens, Allen, & Sheeber, 2010). Self-report on momentary affect of participants.
Attention (state) | From day 1 till day 40, six times a day between 10 am and 8 pm
  A single self-report item assessing momentary attention: "For the last 30 minutes I have had problems concentrating."
Four items from the Situational Motivation Scale (SIMS) | From day 1 till day 40, six times a day between 10 am and 8 pm
  Self-report of participants on momentary intrinsic motivation, identified regulation, external regulation, and amotivation.
Five emotion regulation strategies (Koval, Brose, Pe et al., 2015) | From day 1 till day 40, six times a day between 10 am and 8 pm
  Self-report on momentary emotion regulation strategies of participants.
Three items from the Dutch eating behavior questionnaire (DEBQ) | From day 1 till day 40, six times a day between 10 am and 8 pm
  German version of the DEBQ. Self-report on momentary restrictive, emotional and external eating behaviors of participants.
Three items from the Work related Flow Inventory (WOLF) | From day 1 till day 40, six times a day between 10 am and 8 pm
  Self-report on momentary work flow experience of participants.
Three items from the State Adult Attachment Measure (SAAM) | From day 1 till day 40, six times a day between 10 am and 8 pm
  Self-report on current attachment style of participants.
Three items from the Recovery Experience Questionnaire | From day 1 till day 40, six times a day between 10 am and 8 pm
  Self-report on recovery from work in leisure time of participants.
Self-Control Scale (SCS-KD) | at seven weekly laboratory meetings (day 0, 7, 14, 21, 28, 35 and 42)
  German adaptation of the SCS. Self-report on dispositional self-control of participants.
WHO-Five Well-Being Index | Pre- and post measurement (at day 0 and 42)
  German version of the WHO-5 Well-being index. Self-report on well-being of participants.
Emotion Regulation Questionnaire (ERQ) | Pre- and post measurement (at day 0 and 42)
  German adaptation of the ERQ. Self-report on habitual use of emotion regulation strategies (cognitive reappraisal and expressive suppression) of participants.
Adult Attachment Scale (AAS) | Pre- and post measurement (at day 0 and 42)
  German adaptation of the AAS. Self-report on attachment related attitudes of participants.
Dutch eating behavior questionnaire (DEBQ) | Pre- and post measurement (at day 0 and 42)
  German version of the DEBQ. Self-report on restrictive, emotional and external eating behaviors of participants.
Mindful Attention and Awareness Scale (MAAS) | At weekly laboratory meetings (day 0, 7, 14, 21, 28, 35 and 42)
  German version of the MAAS. Self-report on dispositional mindfulness of participants.
Big Five Inventory (BFI-44) | Pre- and Post measurement (at day 0 and 42)
  German adaptation of the BFI-44. Self-report on personality traits of participants.
Breath counting task (Levinson et al., 2014) | Pre- and Post measurement (at day 0 and 42)
  Behavioral measure of mindfulness.
Brief Symptom Inventory (BSI-18) | Pre- and Post measurement (at day 0 and 42)
  German version of the BSI-18. Self-report on symptoms of somatisation, depression and anxiety of participants.
Kentucky Inventory of Mindfulness Skills (KIMS) | Pre- and Post measurement (at day 0 and 42)
  German version of the KIMS. Self-report on mindfulness skills of participants.

OTHER OUTCOMES:
Toronto Mindfulness Scale (TMS) | At weekly laboratory meetings (day 7, 14, 21, 28, 35)
  Self-report on meditation experiences after breathing meditation.

CONTACTS AND LOCATIONS:
Overall Officials: Mario Wenzel, Dipl. Psych., Principal Investigator — Department of Psychology, Johannes Gutenberg University Mainz; Thomas Kubiak, Prof. Dr., Principal Investigator — Department of Psychology, Johannes Gutenberg University Mainz
Locations (1):
- Department of Psychology, Johannes Gutenberg University Mainz, Mainz, Rhineland-Palatinate, Germany

REFERENCES:
- [Background] Bringmann LF, Vissers N, Wichers M, Geschwind N, Kuppens P, Peeters F, Borsboom D, Tuerlinckx F. A network approach to psychopathology: new insights into clinical longitudinal data. PLoS One. 2013 Apr 4;8(4):e60188. doi: 10.1371/journal.pone.0060188. Print 2013. PMID 23593171
- [Background] Levinson DB, Stoll EL, Kindy SD, Merry HL, Davidson RJ. A mind you can count on: validating breath counting as a behavioral measure of mindfulness. Front Psychol. 2014 Oct 24;5:1202. doi: 10.3389/fpsyg.2014.01202. eCollection 2014. PMID 25386148
- [Background] Kuppens P, Allen NB, Sheeber LB. Emotional inertia and psychological maladjustment. Psychol Sci. 2010 Jul;21(7):984-91. doi: 10.1177/0956797610372634. Epub 2010 May 25. PMID 20501521
- [Background] Koval P, Brose A, Pe ML, Houben M, Erbas Y, Champagne D, Kuppens P. Emotional inertia and external events: The roles of exposure, reactivity, and recovery. Emotion. 2015 Oct;15(5):625-36. doi: 10.1037/emo0000059. Epub 2015 Apr 6. PMID 25844974
- [Background] Russell JA. Core affect and the psychological construction of emotion. Psychol Rev. 2003 Jan;110(1):145-72. doi: 10.1037/0033-295x.110.1.145. PMID 12529060
- [Derived] Rowland Z, Wenzel M, Kubiak T. A mind full of happiness: How mindfulness shapes affect dynamics in daily life. Emotion. 2020 Apr;20(3):436-451. doi: 10.1037/emo0000562. Epub 2018 Dec 20. PMID 30570315
- [Derived] Rowland Z, Wenzel M, Kubiak T. The effects of computer-based mindfulness training on Self-control and Mindfulness within Ambulatorily assessed network Systems across Health-related domains in a healthy student population (SMASH): study protocol for a randomized controlled trial. Trials. 2016 Dec 1;17(1):570. doi: 10.1186/s13063-016-1707-4. PMID 27906104